CLINICAL TRIAL: NCT02376348
Title: Increasing Uptake of Voluntary Medical Male Circumcision Among Men Aged 20-34 Years in Njombe & Tabora Regions, Tanzania: A Cluster Randomised Controlled Trial
Brief Title: Male Circumcision Against HIV Hukomboa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Jhpiego (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mwita Wambura, Researcher, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: GH 005-000513
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: VMMC; Adult males; HIV Prevention; Africa

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Individuals receiving the standard Ministry of Health Package
- Intervention (Experimental): Individuals receiving the targeted demand creation strategy to increase adult men taking up VMMC
  Interventions: Behavioral: A targeted demand creation Activities

INTERVENTIONS:
Behavioral: A targeted demand creation Activities — Sites randomized to the intervention arm will receive all activities in the control arm, plus additional demand-creation communication messages that focus on the non-HIV benefits of VMMC and the voluntary nature of HIV testing prior to VMMC ii) use of already circumcised men from the community as auxiliary peer promoters, iii) separate waiting and group education areas for men aged 20 years and above during service delivery, iv) engagement of female partners in community-based demand creation and education and counselling about wound healing and post-circumcision abstinence.
  Arms: Intervention

SUMMARY:
Tanzania launched a National Strategy for scaling-up voluntary medical male circumcision in 2010, and aims to circumcise 2.8 million males by 2015. In September 2009, Jhpiego's Maternal and Child Health Integrated Program (MCHIP) launched a PEPFAR-funded voluntary medical male circumcision (VMMC) program which has circumcised over 110,000 males in Njombe and Iringa regions by June 2012. In line with the national strategy, the target age for the program was 10-34 years, but 80% of clients were aged 10-19 years. There is an urgent need to increase the proportion of older men (aged 20 years and above) who become circumcised, to have greatest impact on the HIV epidemic.

DETAILED DESCRIPTION:
In order to maintain high client flow in sites, the Iringa service delivery model is flexible in terms of how, where and when services are delivered. Approaches include:

i) Static sites: These sites offer regularly scheduled VMMC services several days a week. Services are offered year round rather than periodically. Volume tends to be low (20-50 clients a week).

ii) Outreach sites: VMMC services are offered periodically at health facilities. A team composed of providers 'borrowed' from other regional health facilities visits the sites for a 2-3 week period and offers VMMC 6 days a week. This is typically a high volume setting, in which 40-120 circumcisions are performed a day, depending on the number of beds which can be set up.

iii) Campaign: Campaigns happen 2-3 times a year, and may include both static and outreach sites. Campaigns are high volume, concerted approaches to VMMC where multiple facilities are running coordinated VMMC service delivery.

These services are complemented by demand creation activities (mass media, interpersonal activities and outreach activities) designed to recruit and motivate new clients, and a text messaging information system which is advertised through radio and other means, providing potential clients advice on where VMMC is offered, the benefits of VMMC, and post-surgery reminders for wound care, follow-up visits and safer sex. The intensity of the demand creation depends on the size of campaign. In general, static sites do not have any demand creation but outreach and campaigns do.

The proposed research will take place at outreach sites; however, the study will not stop on-going VMMC services provided at static sites to young men but rather encourage older males to come as well as young boys. Outreach sites have larger potential client size than static sites because the catchment area round the outreach sites have generally not had access to VMMC in the past and clients show up in large numbers to be served, whereas in static sites, clients trickle through in lower volume. Outreach activities can be scheduled at the convenience of the program. By using outreach activities, the proposed research, can be more easily scheduled into the study's data collection timeframe (compared to campaign sites which are on a highly prescribed schedule).

QUALITATIVE ASSESSMENT FINDINGS In February 2011, Jhpiego co-investigators on this study conducted qualitative research in 3 districtsin Iringa (Iringa Municipality, Njombe and Mafinga), with the aim of understanding men's and women's views on appropriate age for circumcision, perceptions on circumcision, barriers and facilitators to older men seeking circumcision, and seasonality[9]. Identified barriers among older men included shame associated with older men getting circumcised, as it was seen to be an age-inappropriate activity, concerns of older men about their partners being faithful to them during the healing period, concerns about loss of income during the healing period, and concern around erections causing damage to the penis or delay wound healing. The facilitating factors included that circumcised men were seen as cleaner, safer from diseases, and more sexually desirable to women.

Exploration of preferences for service delivery showed that participants had a strong preference for a model in which boys and men were provided separate services. There was also support for all-male service providers to alleviate concerns about embarrassment at having women view/touch the penis and the possibility that an erection could occur during the procedure. There was little support for including female partners accompanying their partners to the facilities. There was a marked preference for the cold season (June-August) for three reasons: fewer farming responsibilities, school being out, and a cold temperature which is perceived to facilitate wound healing.

Based on this research, we anticipate that the targeted VMMC strategy evaluated in this research will include demand-creation strategies using focused informational communication messages for men aged over 20 years, and increased information and education for female partners. Service delivery strategies may include separate services for men versus boys and increasing the role of male service providers. The targeting strategy will be finalised during Study 1, and implemented and evaluated during Study 2.

ELIGIBILITY:
Inclusion Criteria:

Sites

* an outreach VMMC health facility,
* a site selected by Jhpiego for outreach VMMC campaign,
* a site that has not had previous outreach services (to enable the results to be generalizable to future new outreach) or have not had VMMC outreach services in the previous 6 months, and
* physically distant from other potential study sites to minimise contamination (spill over) of activities in the intervention communities into control communities.

The parent sites from different clusters must be at least 20km away from each other, regardless of whether they are randomised to be control or intervention sites.

Clients

1. Uncircumcised males
2. given an informed consent to participate in the study

Exclusion Criteria:

1) Circumcised males

Ages: 10 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10782 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Impact of intervention on proportion of male clients aged 20-34 years (ratio of the geometric mean proportion of clients aged 20-34 years in the 10 intervention facilities versus that in the 10 control facilities) | 5-6 weeks of demand creation activities
  Cluster-level summary methods will be used to assess the impact of the intervention[19]. The primary outcome will be the unadjusted "prevalence ratio", estimated as the .

SECONDARY OUTCOMES:
Comparison of population attending for circumcision with general male population (proportion of males reporting the below risk factors will be compared to proportion of males reporting the same in the 2010 Tanzania Demographic and Health Survey) | 5-6 weeks
  In this study, high risk males will be males reporting two or more partners in the last 12 months; reporting unprotected sex with non-married and non-cohabiting sexual partners and men who agreed on a price and paid anyone in exchange for having sexual intercourse. The proportion of males reporting the above risk factors will be compared to proportion of males reporting the same in the 2010 Tanzania Demographic and Health Survey

CONTACTS AND LOCATIONS:
Locations (2):
- Tanzania (2):
  - Njombe, Njombe
  - Tabora, Tabora